CLINICAL TRIAL: NCT01873534
Title: A Phase 2A, Uncontrolled, Open-labeled Trial to Evaluate the Effect of FMX-8 Treatment for Anemia in Patients With End Stage Renal Disease (ESRD) on Hemodialysis (HD)
Brief Title: A Phase 2A Trial of FMX-8 Treatment for Anemia in Patients With ESRD on Hemodialysis HD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit patients meeting the inclusion criteria
Sponsor: FerruMax Pharmaceuticals, Inc. (Industry)
Collaborators: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FX-C-402
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Anemia of Chronic Disease
Keywords: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FMX-8 (0.5 mg/kg) (Experimental): 0.5 mg/kg FMX-8 IV twice per week for 29 days (9 doses)
  Interventions: Drug: FMX-8
- FMX-8 (5 mg/kg) (Experimental): 5 mg/kg FMX-8 IV twice per week for 29 days (9 doses)
  Interventions: Drug: FMX-8
- FMX-8 (15 mg/kg) (Experimental): 15 mg/kg FMX-8 IV twice per week for 29 days (9 doses)
  Interventions: Drug: FMX-8

INTERVENTIONS:
Drug: FMX-8 — FMX-8 is a fusion protein of the human hemojuvelin (HJV) protein.

SUMMARY:
The trial is an uncontrolled, open-label, parallel group clinical trial. Approximately 10 subjects per dose group in 3 groups will be treated twice weekly for a total of 9 doses, followed by a 4-week observation period. Eligible subjects who have Hgb ≥10.5 g/dL and have stable Hgb levels will start the washout period of one to eight weeks. During the washout period, 30 subjects whose Hgb are < 10.0 will complete the baseline assessment to confirm their eligibility. Eligible subjects will be randomly assigned to one of the 3 cohorts in a 1:1:1 ratio. Subjects will be admitted on the day of the first dose and stay in the clinic overnight for pharmacokinetic (PK) sampling after the first (day 1) and the last dose (day 29). FMX-8 will be administered as 30 min i.v. infusion. After the 29-day treatment period, the trial subjects will be observed for an additional 28 days to allow safety and immunogenicity assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are ≥18 years old
* Diagnosed with ESRD and are stable on hemodialysis for more than 3 months
* Maintained stable Hgb for ≥4 weeks prior to screening
* Two consecutive Hgb values ≥10.5 g/dL within 5 weeks of screening
* Body mass index (BMI) between 18 kg/m2 and 42 kg/m2, inclusive, based upon the latest height and weight
* Ferritin levels ≥100 mg/L or Tsat ≥20% or reticulocyte hemoglobin content (CHr) >25 at screening
* Reasonable clearances on dialysis (KT/V ≥1.0) on two prior determinations within 2.5 months
* Able to provide written informed consent
* Able to understand and follow all trial procedures
* Willing to use contraception as detailed in the protocol

Exclusion Criteria:

* Hgb remains unchanged without erythropoietin (<0.5 g/dL decrease during the 8 week maximum erythropoietin-washout period)
* Receipt of iron infusion after the initiation of erythropoietin washout
* Receipt of red blood cell transfusion within four weeks before screening
* Overt gastrointestinal bleeding or other bleeding episode that required transfusion within 2 months prior to screening
* Infection necessitating antibiotic or anti-viral treatment within a month prior to screening
* Requirement for Coumadin (warfarin), Pradaxa or Xarelto
* Hemoglobinopathies such as homozygous sickle-cell disease or thalassemias of all types
* Active hemolysis or chronic hypoxia
* Active malignant diseases (except non-melanoma skin cancer) or life expectancy less than 6 months
* Chronic, uncontrolled or symptomatic inflammatory disease or non-renal cause of anemia such as rheumatoid arthritis, systemic lupus erythematosus, HIV, or systemic acute infection
* On immunosuppressive therapeutics
* Chronic congestive heart failure (New York Heart Association Class III, IV)
* Significant hypertension (≥90 diastolic) based on a sitting diastolic blood pressure at screening
* Kidney transplant within the past year: patients who are off immunosuppressive agents following a failed transplant are eligible for the trial
* End-stage liver disease
* Known hypersensitivity to recombinant protein therapies
* Female patients who are pregnant or breast feeding
* Previous exposure to FMX-8
* Exposure to Omontys® or Hematide® (peginesatide) anemia treatment within the past 6 months
* Treatment with Aranesp® (darbepoetin alpha) within the past 4 weeks
* Uncontrolled hyperparathyroidism (PTH >750) based upon latest PTH determination within the past 4 months
* Inability to comply with the trial scheduled visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who achieve an increase in Hgb ≥ 1g/dL from the lowest Hgb concentration post erythropoietin-washout or continuing rise in Hgb concentration for two consecutive weeks | Weekly for 8 weeks
Number and Severity of Adverse Events | 8 weeks
Serum FMX-8 levels | Dosing Days 1 and 29
  Serum drug levels (pre-dose, and 25 minutes, 35 minutes, 1, 2, 4, 6, 10, 16 and 24 hrs post-dose) will be used to determine, for each dose, standard pK profiles
Number of Subjects with Positive Serum for Anti-Drug Antibodies | At 36 and 57 days after first dose of FMX-8

SECONDARY OUTCOMES:
Changes in Hgb in each dose group during the treatment and follow-up periods | Weekly for 8 weeks
Proportion of subjects that achieve/maintain an absolute Hgb concentration of ≥ 10.0 g/dL for two consecutive weeks | Weekly for 8 weeks
Time to beginning of steady increase of Hgb (for two consecutive weeks) | Weekly for 8 weeks
Time to Hgb increase ≥1 g/dL | Weekly for 8 weeks
Time to full recovery of Hgb to pre- erythropoietin-washout level | Weekly for 8 weeks
Proportion of subjects needing erythropoietin rescue and length of time to start of rescue therapy | Weekly for 8 weeks
Change of hepcidin and erythropoietin | At weeks 2, 4, 6 and 8 from baseline
Changes in Serum Iron, Tsat and plasma Ferritin | At weeks 2, 4, 6 and 8 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Fang, MD, PhD, Study Chair — FerruMax Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - DaVita Arvada Dialysis Center, Arvada, Colorado
  - DaVita Minneapolis Dialysis Unit, Minneapolis, Minnesota